CLINICAL TRIAL: NCT01176708
Title: The Significance of Intact Liver Innervation for the Glucose and GLP-1 Induced Insulin Secretion
Brief Title: Intact Liver Innervation and Glucose and Glucagon-like Peptide-1 (GLP-1) Induced Insulin Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, MD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Transplant isoglycemia (AP)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; kidney transplanted; glucagon-like peptide-1; insulin secretion; vagotomy
MeSH Terms: interventions — Dipeptidyl Peptidase 4; Vildagliptin; Glucose; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liver transplanted (Experimental): 10 Liver transplanted patients
  Interventions: Drug: dipeptidyl peptidase 4 (DPP4) inhibitor; Other: oral glucose; Other: intravenous glucose
- Kidney transplanted (Experimental): 10 kidney transplanted individuals
  Interventions: Drug: dipeptidyl peptidase 4 (DPP4) inhibitor; Other: oral glucose; Other: intravenous glucose
- Healthy controls (Experimental): 10 healthy controls
  Interventions: Drug: dipeptidyl peptidase 4 (DPP4) inhibitor; Other: oral glucose; Other: intravenous glucose

INTERVENTIONS:
Drug: dipeptidyl peptidase 4 (DPP4) inhibitor — One tablet (50 mg)of DPP4 inhibitor is to be taken 12 and 1 hours before start of the oral glucose tolerance test (50 g glucose and 1.5 g paracetamol dissolved in 300 ml water)on day 3
  Other Names: Galvus
Other: oral glucose — 50 grams glucose dissolved in 300 ml water with 1.5 grams paracetamol
  Other Names: Panodil
Other: intravenous glucose — 1.5 g paracetamol dissolved in 50 ml water is to be ingested orally within the first 2 minutes. Intravenous glucose is supplied in an amount to match the plasma glucose during the oral glucose tolerance test
  Other Names: Panodil

SUMMARY:
The aim of the study is to investigate the significance of intact nerve supply to the liver for the glucagon-like peptide-1 (GLP-1) induced insulin secretion.

The hypothesis is that the effects of GLP-1 is transmitted through the GLP-1 receptor and that these effects involve sensory afferent neurons, probably primarily parasympathetic.

DETAILED DESCRIPTION:
GLP-1 is a potent enterogastron and incretin hormone. It is rapidly inactivated by dipeptidyl peptidase IV so only 10-15% enters the systemic circulation. This has led to the hypothesis that GLP-1 interact locally with afferent sensory nerve fibers.

The aim of this study is to investigate the significance of intact liver innervation for the GLP-1 induced insulin secretion in liver transplanted patients; kidney transplanted control patients matched for immunosuppressive treatment, age, gender and body weight; and ten control persons matched for age, gender and body weight.

The insulin secretion will be evaluated from blood samples that will be analyzed for insulin and c-peptide.

ELIGIBILITY:
Inclusion Criteria:

* normal fasting plasma glucose
* normal hemoglobin
* informed consent

Exclusion Criteria:

* type 1 diabetes mellitus or type 2 diabetes mellitus
* body mass index > 30
* inflammatory bowel disease
* intestinal surgery
* serum creatinine > 250 µM and/or albuminuria
* ALAT > 2 x normal value
* Severe cardiac insufficiency
* in treatment with medicine which cannot be paused for 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
insulin secretion | four hours
  The insulin secretion during a four-hour oral glucose tolerance test (OGTT) and an intravenous isoglycaemic clamp is evaluated

SECONDARY OUTCOMES:
plasma glucose | 20 time points within four hours
  20 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma GLP-1 | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma GIP | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma glucagon | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour
plasma GLP-2 | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour.
plasma PYY | 12 time points within four hours
  12 blood samples will be drawn during the four hours OGTT and intravenous isoglycaemic clamp, most frequently during the first hour

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine F' laboratory, Hellerup, Copenhagen, Denmark